CLINICAL TRIAL: NCT03838861
Title: A Randomised Clinical Trial Testing the Effect of an Individualised and Patient-centred Follow-up Program for Women With Gynaecological Cancer
Brief Title: An Individualised and Patient-centred Follow-up Program for Women With Gynaecological Cancer
Acronym: NEMO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Southern Denmark (Other)
Collaborators: Region of Southern Denmark (Other); Danish Cancer Society (Other)
Responsible Party: Principal Investigator, Stinne Holm Bergholdt, Principal Investigator, University of Southern Denmark
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Stinne1977
Record Dates: First submitted 2019-02-06; First posted 2019-02-12 (Actual); Last update posted 2022-04-22 (Actual); Status verified 2022-04

CONDITIONS: Empowerment, Cervical Cancer, Endometrial Cancer, Follow-up, Nurse-led, PROM
MeSH Terms: conditions — Empowerment; Uterine Cervical Neoplasms; Endometrial Neoplasms; Fetal Membranes, Premature Rupture

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Active Comparator): Standard follow-up in doctors setting
  Interventions: Behavioral: NEMO: NEw MOdel of follow-up
- Intervention (Experimental): Nurse-led follow-up with focus on empowerment and need assessment by use of ePROMS
  Interventions: Behavioral: NEMO: NEw MOdel of follow-up

INTERVENTIONS:
Behavioral: NEMO: NEw MOdel of follow-up — The nurse led model is built upon phone contacts with content and intervals individually planned by the nurse and the patient. The individual contacts will be supported by graphic visualisation of ePROMs in REDCap filled out by the patient before each contact including DGCG's disease specific symptom list and the generic European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30) (24) supplemented with the relevant disease-specific add-on module (25, 26). The sum scores are visualised with colours to indicate severe problems (red), no problems (green) and mild or moderate problems (yellow and orange), respectively. Hence, alarm symptoms and problem areas are clearly presented to the project nurse and changes can be visualised over time enhancing the interpretation. The patient will be given access to own scoring results to obtain an understanding of the meaning of changes in health status.

SUMMARY:
This randomized controlled trial is testing the hypothesis that an individually focused and need-based nurse led follow-up program supported by electronic Patient Reported Outcome Measures for women with gynecological cancer will improve patient's empowerment, quality of life and involvement in the follow-up process besides reducing the patient's fear of cancer recurrence and degree of psychological distress, compared with a doctor led follow-up program. Further, nurse led follow-up by telephone, may reduce resources of the department as well as of the patients.

DETAILED DESCRIPTION:
Background The 2015 release of a new "Follow-up Program for Gynecological Cancers" by the Danish Health Authority (DHA) marked a break with traditional follow-up. The conclusion, derived from a Health Technology Assessment report from 2009 assessing the value of follow up in patients with endometrial and ovarian cancer, was, that regular follow-up visits do not improve survival and may consume unnecessary resources from both patients and health care personnel. As a consequence, a need based program was proposed where the follow-up is planned individually and adjusted according to patient's needs, risks and resources. It was further emphasized that patient's self-care ability should be supported and that access to specialist assessment should be easy available.

The new follow-up program was soon implemented in most national gynecological centers without previous evaluation in a pilot setting and with sparse evidence of benefits and harms. Further, as the recommendations from the DHA were broad, various forms of the model were introduced. Optimally, a national common professional agreement to standardize this transformation should be made. However, there is neither consistency nor sufficient knowledge about the optimal organizational follow-up model for gynecological cancer patients for this to be accomplished.

Internationally, various follow-up models for patients with cancer have been tested over the past decade. In the gynecological setting, evidence of the most optimal organization of follow-up is sparse. In general, studies suggest that follow-up conducted in a nurse or general practitioner setting demonstrate similar survival and recurrence detection rates and similar or slightly better rates of satisfaction and quality of life as compared to follow-up in a conventional setting.

From previous national studies on survivorship in Danish cancer patients it was learned learned that involvement of the general practitioners (GPs) in the follow-up process was not superior, and one in ten cancer patient was not satisfied with the contribution from their GP during the follow-up. Further, studies have shown that socioeconomic status had a significant impact on participation in rehabilitation activities of gynecological cancer patients with cervical and ovarian cancer patients being especially vulnerable. Unmet needs after cancer was found to be significantly associated with lower quality of life emphasizing the importance of need assessment. Preliminary data from a local randomized trial of follow up vs. no follow up in low risk endometrial cancer patients indicate that women report a higher degree of fear of recurrence after cancer treatment if they receive no follow-up as compared to a group receiving conventional follow-up. Hence, results obtained from prior studies on survivorship following gynecological cancer treatment indicate that follow-up to some extent seems needed and emphasize a need to develop new programs that facilitates self-management but at the same time embrace those most vulnerable. Question is how the patients needs are best accommodated with limited resources available. Comprehensive evaluation of effects, benefits and harms are essential before implementation of new initiatives.

This randomized study suggests a strong focus on promotion of cancer patients' self-care ability, in this study conceptualized as empowerment. Empowerment has been described as "a process by which people, organizations, and communities gain mastery over their affairs" and empowerment processes as "processes in which attempts to gain control, obtain needed resources, and critically understand one's social environment are fundamental. The process is empowering if it helps people to develop skills so that they can become independent problem-solvers and decision-makers". Focus on improvement of patient empowerment may thus unify the need for patient involvement, promotion of self-care ability and re-allocate resources to those patients most vulnerable who are often neglected in the follow-up process. Further, by empowering patients to master the consequences of their cancer disease, they may have fewer unmet needs, which may altogether improve quality of life and reduce fear of recurrence.

Use of electronic Patient Reported Outcome Measures (ePROMs) in the follow-up process has in selected populations shown to improve quality of life, reduce emergency room visits and hospitalizations, and improve quality-adjusted survival. Therefore ePROMs are suggested as important elements of future follow-up programs for cancer patients.

By combining nurse-led, needs based and individually planned follow-up, support of patient empowerment to self-manage with use of ePROMS to provide a safe and efficient follow-up program, the extended model of follow-up of the present study may improve patient outcomes and reduce economic as well as human resourses.

Study design Randomized, controlled study. Patients and health care professionals are not blinded, but randomization will be carried out centrally and the allocation sequence is computer-generated with varying block size and is kept unknown for all investigators. In addition, the patient's randomization status will be blinded during data processing and analysis.

The study will be developed, implemented and results will be published in accordance with the CONSORT statement.

Participants and Setting Women with cervical or endometrial cancer who are surgically treated at the Department of Gynecology at Odense University Hospital (OUH) are invited to participate. Women referred to oncological treatment post operative, who do not speak or read Danish, or where consent is unethical, i.e. caused by dementia, are not eligible. Patients will be recruited from 2019-2021.

The project is carried out by project nurses and doctors of the Department of Gynecology at OUH, where inclusion of patients and follow-up are conducted. The department operates 350-400 gynecological cancer patients annually, of which 50-70 with cervical cancer and 160-180 with endometrial cancer. Overall, about 60% (126-150 patients per year) will meet the inclusion criteria.

Patients, who do not wish to participate or for other reasons are not included, are referred to the doctor led follow-up program, which was implemented as the new standard during the autumn of 2017.

The project group consists of clinicians and researchers from the Department of Gynecology at OUH and Clinical Institute, Research Unit for General Practice, and Department of Psychology at University of Southern Denmark. In addition, patient representatives from the Danish "Patient Association of Women with Gynecological Cancer" are invited to give feedback on the proposed intervention, the questionnaires and all patient materials. In addition they will be asked to participate in the interpretation of the study results.

Odense Patient data Explorative Network (OPEN) which is a non-profit research infrastructure of OUH and University of Southern Denmark, contribute to the management of the questionnaires and data collection by using the Research Electronic Data Capture (REDCap) technology. Further, OPEN provides data management assistance and statistical support.

Study plan In the present study an innovative model is tested where specialized nurses handle the follow-up of endometrial and cervical cancer patients in the intervention group. The model is based on telephone consultations and developed to ensure timely identification of alarm symptoms and potential needs and support of the patient's empowerment to manage life after cancer.

Until the intervention baseline at 4 months post operative, all patients receive the same follow-up. Hence, before randomization, all patients are offered a follow-up consultation with a nurse 4 weeks post operative, where a need assessment is conducted using the "Preparatory Form for the patient" as described by the Region of Southern Denmark in their "Guide to need assessment of patients with cancer". Further, a disease specific list of alarm symptoms prepared by working groups of the Danish Gynecological Cancer Group (DGCG) is reviewed with the patient. The patient is carefully instructed to be aware of and contact the department in case of symptoms from the list as they may indicate recurrence, and that access to clinical examination is available and provided when needed.

All patients are eventually offered a follow-up consultation with a doctor 4 months post operative, where a clinical assessment is performed and the Preparatory Form and symptom list are reviewed as part of the needs assessment. If the patient meets the inclusion criteria, she is asked to participate in the study and is randomized if consent is obtained. The randomization status is immediately revealed. For control group patients a new appointment with the doctor is arranged if needed, and for patients in the intervention group a telephone follow-up with the attending nurse is arranged.

ELIGIBILITY:
Inclusion Criteria:

* No adjuvant therapy after surgery
* Speak and write Danish
* Mentally capable to adapt to intervention

Exclusion Criteria:

* Indication for adjuvant therapy after primary surgical treatment

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Female genital cancer patients
Enrollment: 200 (Estimated)
Dates: Start 2019-03-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2025-01-28 (Estimated)

PRIMARY OUTCOMES:
Patient Empowerment using the Health Education Impact Questionnaire (HEI-Q) | Change from baseline (3 months post operative) to 12 months post operative.
  The primary outcome is measured as change of the skill and technique acquisition subscale score of the HEI-Q from baseline to 12 months post operative. Questionnaires are administered at 3 (baseline), 12, 24 and 36 months after surgery, respectively. Change from baseline to 24 and 36 months post operative are considered as secondary outcomes.

SECONDARY OUTCOMES:
Patient Empowerment using the Health Education Impact Questionnaire (HEI-Q) | Questionnaires are administered at 3 (baseline), 12, 24 and 36 months after surgery, respectively
  Change in other subscales of the HEI-Q from baseline to 12, 24 and 36 months post operative
Fear of cancer recurrence using the Fear of Cancer Recurrence Inventory (FCRI) | Questionnaires are administered at 3 (baseline), 12, 24 and 36 months after surgery, respectively
  Change in fear of cancer recurrence from baseline to 12, 24 and 36 months respectively.
Health related quality of life using the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30) | Questionnaires are administered at 3 (baseline), 12, 24 and 36 months after surgery, respectively
  Change in Global Health Status and other subscales of the C30 questionnaire from baseline to 12, 24 and 36 months respectively.
Cancer type specific quality of life using the EORTC Endometrial Cancer Module (EORTC QLQ-EN24) | Questionnaires are administered at 3 (baseline), 12, 24 and 36 months after surgery, respectively
  Change from baseline to 12, 24 and 36 months respectively.
Cancer type specific quality of life using the EORTC Cervical Cancer Module (EORTC QLQ-CX24) | Questionnaires are administered at 3 (baseline), 12, 24 and 36 months after surgery, respectively
  Change from baseline to 12, 24 and 36 months respectively.
Health Status using the EuroQol five-Dimensional (EQ5D) measure | Questionnaires are administered at 3 (baseline), 12, 24 and 36 months after surgery, respectively
  Change from baseline to 12, 24 and 36 months respectively.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Gynecology, Odense University Hospital, Odense, Region Syddanmark, Denmark

REFERENCES:
- [Derived] Bergholdt SH, Hansen DG, Johnsen AT, Boman BS, Jensen PT. A NEw MOdel of individualized and patient-centered follow-up for women with gynecological cancer (the NEMO study)-protocol and rationale of a randomized clinical trial. Trials. 2023 Feb 1;24(1):74. doi: 10.1186/s13063-022-07022-0. PMID 36726187